CLINICAL TRIAL: NCT00327496
Title: Cytotoxicity Induced by Tumor Lysate Pulsed Dendritic Cells Against Autologous Hepatocellular Carcinoma Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mackay Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMH-I-S-166
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2005-06

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

INTERVENTIONS:
Biological: DC vaccine

SUMMARY:
Hepatoma ranks the first on the cancer mortality list in Taiwan, and there are currently no other effective treatment options for advanced HCC. Therefore, alternative medical intervention is needed to improve the survival and quality of life of these patients. Dendritic cells are the most potent type of antigen presenting cells in the human body, and are involved in the regulation of both innate and adoptive immune responses. If we use matured antigen presenting cells pulsed in vitro with appropriate tumor associated antigens under optimal activation conditions. It is anticipated that such treatment might generate or reactivate a cytotoxic T lymphocyte response against tumor cells and thereby inhibit tumor growth.

Although there are excited results of tumor vaccine in animal models but successful clinical tries are rare. There are still some problems needed to be resolved such as immune deficiency of the cancer patients or the defect of T cell receptors or the problems of tumor escape. There are complex compositions in tumor cells to be a tumor antigen that will influence the efficacy of tumor vaccine, so we are going to use tumor lysate to be a tumor antigen.

In this study, the generation of dendritic cells from the patient's peripheral blood will use rhGM-CSF and rhIL-4 as stimulating factors, and matured dendritic cells will pulse with tumor lysate, the ex vivo T cell cytotoxicity for the primary tumor cell will be test. We hope to cooperate with basic study group in our hospital to do more ex vivo tests and clinical trials in the future.

DETAILED DESCRIPTION:
Hepatoma ranks the first two of the cancer mortality list in Taiwan, and there are currently no effective treatment options for advanced HCC. Therefore, novel medical intervention is needed to improve the survival and quality of life of these patients. Dendritic cells are the most potent type of antigen presenting cells in the human body, and are involved in the regulation of both innate and adoptive immune responses. It is assumed that matured antigen presenting cells pulsed in vitro with appropriate tumor associated antigens under optimal activation conditions might generate or activate a cytotoxic T lymphocyte response against tumor cells and thereby inhibit tumor growth(1,2).

Although there are exciting results of tumor vaccine in animal models but successful clinical tries are lacking. There are some problems needed to be resolved such as immune deficiency of the cancer patients, defect of T cell receptors or the immune evasion of tumor. The efficacy of tumor vaccine is mainly affected by both the heterogenicity of tumor cells and complexity of tumor antigens. Tumor lysates which include multiple antigens, are supposed to be a good source of tumor antigens(3-7). The purpose of this study is to investigate the ability of autologous peripheral blood monocyte-derived dendritic cells (DCs) from hepatoma patients pulsed with autologous tumor lysate to elicit T cells cytotoxicity against hepatoma cells ex vivo. We plan to do HCC primary culture and DCs are derived from peripheral blood monocytes by triggering differentiation with recombinant human granulocyte macrophage colony stimulating factor (rhGM-CSF) and interleukin-4 (rhIL-4) to immature DCs. Immature DCs will be pulsed with autologous hepatoma cell lysates and matured by using a cytokine cocktail. Surface molecule expression on DCs will be analysed by flow cytometry. The ability of the pulsed DCs to stimulate autologous T cell proliferation will be assessed by using carboxyfluorescein diacetate, succinimidyl ester (CFSE) staining. The cytotoxicity of DC-stimulated T cells against primarily cultured hepatoma cells will be estimated by using trypan blue exclusion test. The purpose is to investigate the ability of autologous peripheral blood monocyte-derived dendritic cells (DCs) from hepatoma patients pulsed with autologous tumor lysate to elicit T cells cytotoxicity against hepatoma cells ex vivo.

Reference

1. Liu KJ, Wang CC, Chen LT, Cheng AL, Lin DT, Wu YC, Yu WL, Hung YM, Yang HY, Juang SH, Whang-Peng J. Generation of carcinoembryonic antigen (CEA)-specific T-cell responses in HLA-A*0201 and HLA-A*2402 late-stage colorectal cancer patients after vaccination with dendritic cells loaded with CEA peptides. Clin Cancer Res. 2004 Apr 15;10(8):2645-51. PMID: 15102666
2. Chan RC, Pang XW, Wang YD, Chen WF, Xie Y. Transduction of dendritic cells with recombinant adenovirus encoding HCA661 activates autologous cytotoxic T lymphocytes to target hepatoma cells. Br J Cancer. 2004 Apr 19;90(8):1636-43. PMID: 15083197
3. Iwashita Y, Tahara K, Goto S, Sasaki A, Kai S, Seike M, Chen CL, Kawano K, Kitano S. A phase I study of autologous dendritic cell-based immunotherapy for patients with unresectable primary liver cancer. Cancer Immunol Immunother. 2003 Mar;52(3):155-61. Epub 2003 Feb 06. PMID: 12649744
4. Ladhams A, Schmidt C, Sing G, Butterworth L, Fielding G, Tesar P, Strong R, Leggett B, Powell L, Maddern G, Ellem K, Cooksley G. Treatment of non-resectable hepatocellular carcinoma with autologous tumor-pulsed dendritic cells. J Gastroenterol Hepatol. 2002 Aug;17(8):889-96. PMID: 12164965
5. Parajuli P, Sloan AE. Dendritic cell-based immunotherapy of malignant gliomas. Cancer Invest. 2004;22(3):405-16. PMID: 15493362
6. Song SY, Kim HS. Strategies to improve dendritic cell-based immunotherapy against cancer. Yonsei Med J. 2004 Jun 30;45 Suppl:48-52. PMID: 15250050
7. Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. PMID: 15122249

ELIGIBILITY:
Inclusion Criteria:

* Hepatoma patients indicated for operation

Exclusion Criteria:

* With major systemic disease including other cancer or coagulopathy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-06; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chung Lin, MD, Principal Investigator — Division of Gastroenterology, Mackay Memorial Hospital